CLINICAL TRIAL: NCT02293967
Title: An Open-label, Mass Balance Study to Investigate the Absorption, Metabolism and Excretion of [14C] MT-1303 After a Single Oral Dose to Healthy Male Subjects.
Brief Title: Mass Balance Study of MT-1303
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT-1303-E11
Record Dates: First submitted 2014-11-14; First posted 2014-11-19 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Relapsing-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — amiselimod

ARMS (1):
- MT-1303 (Experimental): [14C] MT-1303 after a single oral dose
  Interventions: Drug: MT-1303

INTERVENTIONS:
Drug: MT-1303

SUMMARY:
The purpose of this study is to investigate the absorption, metabolism and excretion of MT-1303 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male aged 30 to 65 at Screening.
* Body weight of ≥60 kg, and a BMI ranging from 18.0 to 32.0 kg/m2 at Screening and Day -1.
* Normal or not clinically significant ECG as defined by a HR between 50 and 100 bpm inclusive at Screening, Day -1 and pre-dose.
* Vital signs within the following ranges at Screening and Day -1,Body temperature: 35.0 to 37.5 °C,SBP: 90 to 140 mmHg,DBP: 50 to 90 mmHg.
* Regular daily bowel movements.

Exclusion Criteria:

* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study.
* Previous medical history of tuberculosis, or in the opinion of the Investigator, a recurrent medical history of cold sores, pharyngitis, urinary tract infection, diarrhoea/dysentery, chest infections or fungal infections.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardise the subject in case or participation in the study. The investigator should be guided by evidence of any of the following:

  * history of inflammatory bowel syndrome,gastritis, ulcers, gastrointestinal or rectal bleeding;
  * history of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Total radioactivity in urine and faeces | up to 10 weeks

SECONDARY OUTCOMES:
PK of total radioactivity in plasma | up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, Principal Investigator — Quotient Clinical
Locations (1):
- Investigational site, Ruddington, Nottingham, United Kingdom

REFERENCES:
- [Derived] Kifuji T, Inoue S, Furukawa M, Perez Madera B, Goto T, Kumagai H, Mair SJ, Kawaguchi A. Absorption, disposition and metabolic pathway of amiselimod (MT-1303) in healthy volunteers in a mass balance study. Xenobiotica. 2019 Sep;49(9):1033-1043. doi: 10.1080/00498254.2018.1525508. Epub 2018 Dec 21. PMID 30231665